CLINICAL TRIAL: NCT00939367
Title: Randomized, Two Period Crossover Studies in Fed Healthy, Normal Subjects to Compare the Single Dose Bioavailability of Torrent's Zolpidem Tartrate Tablets 10 mg and Sanofi-Synthelabo's Ambien® 10 mg Tablets
Brief Title: Bioequivalence Study of Torrent Pharmaceutical Ltd.'s Zolpidem Tartrate Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: US/05/004
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — Zolpidem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Torrent's Zolpidem TartrateTablets 10 mg
  Interventions: Drug: Zolpidem Tartrate Tablets 10 mg
- Reference (Active Comparator): Sanofi-Synthelabo Inc's Ambient® Tablets 10 mg
  Interventions: Drug: 'Sanofi-Synthelabo Inc's Ambien® Tablets 10 mg

INTERVENTIONS:
Drug: Zolpidem Tartrate Tablets 10 mg
  Arms: Test
Drug: 'Sanofi-Synthelabo Inc's Ambien® Tablets 10 mg
  Arms: Reference

SUMMARY:
Subjects to compare the single dose bioavailability of Torrent's Zolpidem Tartrate Tablets 10mg and Ambien® Tablets 10 mg of Sanofi-Synthelabo Inc.

DETAILED DESCRIPTION:
An Open Label, Randomized, 2-period, 2- Treatment, 2-Sequence, Crossover, Single-dose Bioequivalence Study of Zolpidem Tartrate Tablets containing Zolpidem Tartrate 10 mg ( Test Formulation, Torrent Pharmaceutical Ltd., India) Versus Ambien® Tablets 10 mg containing Zolpidem Tartrate 10 mg (Reference , Sanofi-Synthelabo Inc) in Healthy Human Volunteers Under Fed Condition.

ELIGIBILITY:
Inclusion Criteria:

* The subjects who qualify for the study should meet the following inclusion criteria.

  1. Male and female subjects in the range of 18 - 45 years of age.
  2. Subjects having Body Mass Index (BMI) in a range of 18.5 to 24.9.
  3. Subjects with normal findings as determined by baseline history, physical examination and vital signs (blood pressure, pulse rate, respiration rate and body temperature)
  4. Subjects with normal findings as determined by hematological tests, serum chemistry, urine analysis, ECG and X-ray.
  5. Willingness to follow the protocol requirement as evidenced by written, informed consent.
  6. Agreeing to, not using any medication prescription and over the counter medicines including vitamins and minerals for 14 days prior to study and during the course of the study.
  7. No history or presence of significant alcoholism or drug abuse in the past one year.
  8. Non-smokers, ex smokers and light smokers will be included. " Light smokers are defined as someone smoking 10 cigarettes or less per day, ex smokers as someone who completely stopped smoking for at least 3 months.

Exclusion Criteria:

* The subjects who qualify for the study should not meet the following exclusion criteria:

  1. Requiring medication for any ailment including enzyme-modifying drugs in the previous 28 days, before day1.
  2. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
  3. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic diseases.
  4. Participation in a clinical drug study or bioequivalence study 90 days prior to present study.
  5. History of malignancy or other serious diseases.
  6. Refusal to abstain from food for at least ten (10) hours prior to High Fat Breakfast and for additional four (4) hours post dose during each study period.
  7. Refusal to abstain from water for at least one (1) hour prior to study drug administration on each study period and for at least two (2) additional hours, post dosing.
  8. Any contraindication to blood sampling.
  9. Use of xanthine-containing beverages or food and grapefruit juice for 48 hours prior to each drug dose.
  10. Blood donation 90 days prior to the commencement of the study.
  11. Subjects with positive HIV tests, HbsAg or Hepatitis-C tests.
  12. Known history of hypersensitivity to zolpidem Tartrate or to any of the inactive ingredients in the formulation.
  13. Refusal to abstain from smoking or consumption of tobacco products 24 hours before dosing until last sample collection of each period.
  14. Pregnant and lactating women.
  15. Use of prescription medication within 14 days prior to administration of study medication or over the counter products (including natural food supplements,vitamins, garlic as a supplement) within 14 days prior to administration of study medication, except for topical products without systemic absorption.
  16. Female subjects whose menstruation cycle coincides with the study periods.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-02-24 (Actual); Primary Completion 2007-05-02 (Actual); Study Completion 2007-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Accutest Research Laboratories Pvt. Ltd., Mumbai, Maharashtra, India

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: healthy, normal subjects
Groups:
- Torrent's Zolpidem First, Then Ambien: For period one - on the morning of Day 1 subjects received Torrent's Zolpidem 10 mg.
  Followed by a 7 day washout period.
  For period two - on the morning of Day 1 subjects received the reference formulation, Ambien 10 mg.
- Ambien First, Then Torrent's Zolpidem: For period one - on the morning of Day 1 subjects received the reference formulation, Ambien 10 mg
  Followed by a 7 day washout period.
  For period two - on the morning of Day 1 subjects received the test formulation, Torrent's Zolpidem 10 mg.
Period: First Intervention
Arm/Group | Torrent's Zolpidem First, Then Ambien | Ambien First, Then Torrent's Zolpidem
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Torrent's Zolpidem First, Then Ambien | Ambien First, Then Torrent's Zolpidem
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Torrent's Zolpidem Tartrate Tablets 10 mg and Ambien® 10mg tablets
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (7.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Region of Enrollment [Number; unit: participants]
  India | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma
Time Frame: plasma samples were obtained from blood drawn at 0 (within 60 minutes prior to dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 20 and 24 hours (18 samples) after administration of the dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Experimental: Torrent's Zolpidem Tartrate Tablets 10 mg
- Active Comparator: Ambien® 10mg tablets
Arm/Group | Experimental | Active Comparator
Number analyzed (Participants) | 30 | 30
ng/mL | 130.58 (40.61) | 124.53 (37.48)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | Experimental | Active Comparator
Number analyzed (Participants) | 30 | 30
ng.hr/mL | 734.29 (416.53) | 705.45 (356.65)

3. Primary Outcome: The Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity AUC(0-∞)
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | Experimental | Active Comparator
Number analyzed (Participants) | 30 | 30
ng.hr/mL | 776.65 (484.20) | 734.01 (384.90)

ADVERSE EVENTS:
Arm/Group | Experimental | Active Comparator
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=30) | Active Comparator (N=30)
Regurgitation of water and food content (General disorders) | 2 (2) | 1
Giddiness (General disorders) | 1 (1) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other